CLINICAL TRIAL: NCT01922492
Title: Effect of Islet Autotransplantation Compared to Oral Antidiabetic Drug in Partially Pancreatectomized Patients Due to Benign Pancreatic Neoplasm.
Brief Title: Effect of Islet Autotransplantation Compared to Oral Antidiabetic Drug.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Novartis (Industry)
Responsible Party: Principal Investigator, Kyong Soo Park, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHUH_AIT_1
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Partial Pancreatectomy Due to Benign Pancreatic Neoplasm
Keywords: autologous islet transplantation; partial pancreatectomy; pancreatogenic diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous islet transplantation (Experimental): Autologous islet transplantation arm: autologous islet transplantation
  Interventions: Procedure: Autologous islet transplantation
- Oral anti-diabetic drugs (Active Comparator): Metformin (starting from 500mg qd with dose adjustment thereafter) with or without vildagliptin (starting from 50mg qd with dose adjustment thereafter)
  Interventions: Drug: Oral anti-diabetic drugs

INTERVENTIONS:
Procedure: Autologous islet transplantation — Islet was isolated from the normal part of resected pancreas with modified Ricordi method.
  After purification, the islets were infused into the liver through percutaneous transhepatic portal vein catheterization.
  Arms: Autologous islet transplantation
Drug: Oral anti-diabetic drugs — * Metformin on the diagnosis of postoperative diabetes mellitus. Starting dose of 500mg per day and dose adjustment as needed to control blood glucose.
  * Vildagliptin added on the insufficient glycemic control with monotherapy. Starting dose of 50mg per day and dose adjustment as needed to control blood glucose.
  Arms: Oral anti-diabetic drugs

SUMMARY:
* Effects of autologous islet transplantation were compared to those of oral anti-diabetic drugs after distal pancreatectomy.
* The primary interest is a insulin-secretory function after the surgery in two intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent distal pancreatectomy for pathologic diagnosis of pancreatic mass

Exclusion Criteria:

* Prior history of diabetes mellitus
* Patients whose fasting, post-load (75g OGTT) glucose or HbA1c level meet ADA diagnostic criteria
* Patients who refused to participate the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes of insulin secretory function | preop., 1 week and 1 month postop., and every 3 months after the surgery until 5 year postop.
  Insulin secretion was evaluated by calculating insulinogenic index (Δ insulin30min (μIU/ml)/Δglucose30min (mmol/L) during 75g-OGTT) and homeostasis model assessment for beta cell function (HOMA-B).

SECONDARY OUTCOMES:
Changes of glucose tolerance | preop., 1 week and 1 month postop., and every 3 months after the surgery until 5 year postop.
  Glucose tolerance was evaluated by HbA1c (%), 1,5-anhydroglucitol (ug/ml), and area under the curve of glucose (75g OGTT, mg/dl*min).
Incidence of postoperative diabetes mellitus | preop., 1 week and 1 month postop., and every 3 months after the surgery until 5 year postop.
Changes of insulin resistance | preop., 1 week and 1 month postop., and every 3 months after the surgery until 5 year postop.
  Insulin resistance was evaluated by homeostasis model assessment for insulin resistance (HOMA-IR).
Adverse effects | preop., 1 week and 1 month postop., and every 3 months after the surgery until 5 year postop.

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Soo Park, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoon JW, Jung HS, Jang JY, Kim MJ, Kim JH, Ohn JH, Kim JH, Lee HM, Kim HC, Lee KB, Choi SA, Kim SW, Park KS. Improved Insulin Secretion by Autologous Islet Transplantation, Compared to Oral Antidiabetic Agents, After Distal Pancreatectomy. Cell Transplant. 2015;24(8):1615-26. doi: 10.3727/096368914X682440. Epub 2014 Jun 27. PMID 24978858